CLINICAL TRIAL: NCT02235714
Title: Exhaled Breath Condensate Biomarkers of Inflammation in Individuals With Chronic Cervical Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Miroslav Radulovic, M.D., Staff Physician, James J. Peters Veterans Affairs Medical Center
Other Study IDs: RAD-09-031
Record Dates: First submitted 2012-12-05; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Tetraplegia; Asthma
Keywords: Airway inflammation; Tetraplegia; Asthma; Exhaled breath condensate; Spirometry; Pulmonary Function Testing
MeSH Terms: conditions — Quadriplegia; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled Breath Condensate Blood Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Tetraplegia: Individuals with chronic tetraplegia
- Asthma: Individuals with mild asthma
- Able-bodied controls: Age matched able-bodied (AB) controls with no history of lung disease

SUMMARY:
The purpose of this study is to obtain markers of airway inflammation from the exhaled breath condensate (the moisture in exhaled air) for comparison to blood based markers. These markers will be compared in tetraplegic, asthmatic and able-bodied control groups. Additionally, lung function testing will be performed, and the associations between breath condensate and blood markers and pulmonary function explored between groups.

DETAILED DESCRIPTION:
The predominant mechanism for pulmonary dysfunction in individuals with chronic tetraplegia is respiratory muscle paralysis. This leads to inadequate ventilation and inability to clear secretions placing these patients at a greater risk for the development of respiratory complications. Furthermore, individuals with chronic tetraplegia exhibit baseline increases in airway tone (bronchoconstriction), restoration of normal airway caliber following bronchodilator administration, and non-specific airway hyperresponsiveness (AHR) following inhalation of methacholine, histamine, an aerosolized distilled water. These findings in persons with spinal cord injury (SCI) represent pulmonary features commonly seen in individuals with asthma. Alternatively, airway inflammation may play a role in the obstructive physiology observed in individuals with tetraplegia. In this population, identification of cellular inflammation would confirm the presence of underlying inflammation with a sputum induction. However, this method is hard to perform due to an impaired cough.

The emerging field of exhaled breath condensate (EBC) biomarkers of inflammation offers a non-invasive technique to define the presence of, and potentially address the contributing factors of airway inflammation in the respiratory tract of individuals with tetraplegia. It is thought that EBC composition reflects biochemical changes of airway lining fluid. EBC contains a large number of mediators, including adenosine, ammonia, hydrogen peroxide (H2O2), isoprostanes, leukotrienes, prostanoids, peptides and cytokines. Looking at exhaled breath profiles of various biomarkers may be used to differentiate their different pathophysiological mechanism of inflammation. In addition, measurements of some chemokines (TNF-ά, interleukin (IL)-6) and inflammatory biomarkers (LTB4) in EBC and blood simultaneously may help differentiate the degree of local vs. systemic inflammation. Understanding the underlying mechanisms involved in pulmonary dysfunction observed in persons with chronic cervical SCI may identify treatment options, such as use of inhaled steroids. This approach would be expected to ultimately improve quality of life in affected individuals, decreasing the rate of re-hospitalizations due to respiratory complications and the socioeconomic burden placed on these with SCI and the health care system.

ELIGIBILITY:
Inclusion Criteria:

(1) 18 to 65 years old.

Groups:

1. Chronic stable tetraplegia (duration of injury > 1 year) matched for age, gender, and BMI with healthy control subjects, and clinically stable mild asthmatic subjects. The subjects approached will have already consented to, or be actively participating in "Effects of Nitric Oxide Synthase Inhibitor on Levels of Exhaled NO and Airway Tone in Subjects with Chronic Cervical Spinal Cord Injury" study.
2. Clinically stable mild asthmatic subjects (as defined by NIH asthma guidelines) [51].
3. Healthy able-bodied individuals.

Exclusion criteria (all subjects):

1. Smoking, active or history of smoking during life time.
2. More than mild airflow obstruction as per spirometric indices,
3. Active respiratory disease,
4. Medications known to affect the respiratory system,
5. Pregnancy and
6. Lack of mental capacity to give informed consent.
7. No history of asthma diagnosis during lifetime (able bodied and tetraplegia groups), or recent (within 3 months) respiratory infection for all groups.
8. Receiving medications known to alter airway caliber.

Exclusion Criteria (specific to Asthmatic subjects):

1. Moderate to severe airflow obstruction as per spirometric indices,
2. Testing within 48 hours of last administration of long-acting inhaled bronchodilator medication,
3. Testing within 7 days of last administration of inhaled or oral corticosteroid medication,
4. Testing within 24 hours since last administration of leukotriene modifiers and
5. Testing within 8 hours of last administration of a short-acting inhaled bronchodilator medications

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Chronic stable tetraplegia (duration of injury > 1 year) matched for age, gender, and BMI with healthy control subjects, and clinically stable mild asthmatic subjects. The subjects approached will have already consented to, or be actively participating in "Effects of Nitric Oxide Synthase Inhibitor on Levels of Exhaled NO and Airway Tone in Subjects with Chronic Cervical Spinal Cord Injury" study.
  2. Clinically stable mild asthmatic subjects (as defined by NIH asthma guidelines) [51].
  3. Healthy able-bodied individuals.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Levels of inflammatory biomarkers | Baseline
  To compare the levels of inflammatory biomarkers in exhaled breath condensate (breath condensate acidity, 8-isoprostane, LTB4, prostaglandin E2, IL-6, TNF-ά in individuals with tetraplegia to that of matched control subjects diagnosed with asthma (positive control) and healthy able-bodied individuals (negative controls).

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Radulovic, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States